CLINICAL TRIAL: NCT01897428
Title: Clinical Trial to Evaluate Pharmacokinetic Characteristics of Belion in Healthy Subjects
Brief Title: PK Comparisons of Bepotastine Besilate 10 mg and Bepotastine Salicylate 9.64 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Ji-Young Park, Associate Professor of Clinical Pharmacology, Korea University Anam Hospital
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HL-BPT-101
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2011-03

CONDITIONS: Allergic Rhinitis; Urticaria; Pruritus
MeSH Terms: conditions — Rhinitis, Allergic; Urticaria; Pruritus | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference arm (Active Comparator): Treated with Reference (bepotastine besilate 10 mg)
  Interventions: Drug: Reference-bepotastine besilate 10 mg
- Test arm (Experimental): Treated with Test (bepotastine salicylate 9.64 mg)
  Interventions: Drug: Test-Bepotastine salicylate 9.64 mg

INTERVENTIONS:
Drug: Test-Bepotastine salicylate 9.64 mg
  Other Names: Berion; Manufactured by Hanlim Pharm. Co., Ltd, Seoul, Korea
  Arms: Test arm
Drug: Reference-bepotastine besilate 10 mg
  Other Names: Tarion; Manufactured by Dong-A Pharm. Co., Ltd, Seoul, Korea
  Arms: Reference arm

SUMMARY:
To compare the relative bioavailability and pharmacokinetic characteristics of a newly developed bepotastine formulation, bepotastine salicylate, with a conventional formulation, bepotastine besilate, in healthy subjects with a single dose, randomized, open-label, 2-sequence -2period crossover study.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged between 20 and 45 years
* Body weight > 50 kg (in case of female > 45 kg) with BMI between 18 and 29 kg/m2
* Signed and dated informed consent form which meets all criteria of current FDA and KFDA regulations

Exclusion Criteria:

* subjects with acute conditions.
* presence of history affecting ADME
* Clinically significant history or current evidence of a hepatic, renal, gastrointestinal, or hematologic abnormality
* Hepatitis B, hepatitis C, or HIV infection revealed on the laboratory findings
* Any other acute or chronic disease
* A history of hypersensitivity to bepotastine
* A history of alcohol or drug abuse
* Participation in another clinical trial within 2 months
* smoked >10 cigarettes daily
* consumption over 5 glasses daily of beverages containing xanthine derivatives
* use of any medication having the potential to affect the study results within 10 days before the start of the study.
* medication of the inhibitors or inducers of DME including barbiturates within 1 month
* one of abnormal lab findings as like

  * c. AST/ALT > UNL (upper normal limit) x 1.5
  * Total bilirubin > UNL x 1.5

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
bepotastine pharmacokinetics: peak plasma concentrations (Cmax) | 24 hr
Bepotastine Pharmacokinetics: Area under the time vs. plasma concentration curve from 0 to 24 hr(AUCall) | 24 hr
Bepotastine Pharmacokinetics: Area under the time vs. plasma concentration curve from 0 to infinity(AUCinf) | 24 hr

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Clinical Pharmacology & Toxicology, Anam Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim KA, Park JY. Pharmacokinetic comparisons of bepotastine besilate and bepotastine salicylate in healthy subjects. Clin Drug Investig. 2013 Dec;33(12):913-9. doi: 10.1007/s40261-013-0140-7. PMID 24105252